CLINICAL TRIAL: NCT07316244
Title: Pattern of Microbial Keratitis in Assiut University Hospital
Status: Not yet recruiting | Type: Observational
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Liza Mamdouh, Ophthalmology Resident doctor, Assiut University
Other Study IDs: Pattern Mk in A.U.H
Record Dates: First submitted 2025-12-16; First posted 2026-01-05 (Actual); Last update posted 2026-01-05 (Actual); Status verified 2025-12

CONDITIONS: Keratitis; Microbial Keratitis
Keywords: Mk
MeSH Terms: conditions — Keratitis | interventions — Sensitivity and Specificity

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: corneal scraping including direct smear, culture and sensitivity — corneal scraping including direct smear, culture and sensitivity

SUMMARY:
The aim of the study is to explore the epidemiology, including risk factors, causative microorganisms, complications and clinical outcomes of microbial keratitis among patients attending cornea clinic at Assiut University Hospital.

DETAILED DESCRIPTION:
Microbial keratitis (MK) is a potentially-serious, sight-threatening infection that may cause significant visual impairment or even blindness if not diagnosed and treated promptly.It can be caused by a range of pathogens including bacteria (Pseudomonas aeruginosa, Staphylococcus aureus, and Streptococcus pneumoniae), viruses(herpes viruses), parasites (e.g., Acanthamoeba), and fungi (yeasts, and filaments).

Bacterial keratitis (BK) is the most common cause of microbial keratitis Incidence, risk factors and impact of disease, vary widely according to region, access to health care, socioeconomic and environmental factors, predisposing conditions and causative organisms.The frequency and severity of keratitis are significantly higher in low-income countries.

The history of contact lens (CL) wear, ocular trauma, ocular surface disease (e.g. blepharitis, and dry eye), and systemic diseases (diabetes, and rheumatoid arthritis) are common risk factors associated with MK.

Early treatment reduces the risk of corneal scarring, vascularization, or perforation.Treatment with different anti-microbial agents depend on the presenting clinical picture, initiated with broad spectrum empirical antibiotics in suspected bacterial keratitis, prior to targeted treatment guided by corneal scraping for gram-stain, culture and sensitivity.

The diagnosis of MK is made on the clinical basis together with microbiological evaluation. The microbiological profile of microbial keratitis has shown great differences worldwide. Due to the continuous shifting in microbiological profile and antibiotics resistance profiles reported in several studies, microbiological investigations and antibiotic susceptibility are mandatory to provide an effective treatment.

ELIGIBILITY:
Inclusion Criteria:

* All cases presented with Microbial keratitis at cornea clinic , Assiut university hospital during the study period.

Exclusion Criteria:

* Non-microbial keratitis including Moorens ulcers, chemical burns, and Shield ulcers.

Sex: All
Age Groups: Child, Adult, Older Adult
Study Population: 1. Full history taking: age, gender, residency ( urbn or rural ), literacy, present or past medical and surgical histories
  2. Full ophthalmological examination,visual acuity at presentation and after healing.
  3. Slit-lamp biomicroscopy
  3. outcome of corneal scraping including direct smear, culture and sensitivity
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2026-01 (Estimated); Primary Completion 2026-12 (Estimated); Study Completion 2027-03 (Estimated)

PRIMARY OUTCOMES:
pattern of microbial keratitis in Assiut university hospital. | At initial presentation ( baseline)
  Identification of different causative microbial agents of microbial keratitis among patients presenting to Assiut University Hospital.